CLINICAL TRIAL: NCT02014714
Title: Randomized Comparison Study of Single Dose Morphine and Fentanyl Added to Intrathecal Mixture on Orthopedics Patients With Undiagnosed Obstructive Sleep Apnea
Brief Title: Single Dose Morphine and Fentanyl Added to Intrathecal Mixture on Orthopedics Patients With Undiagnosed Obstructive Sleep Apnea
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201311-0466
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Obstructive Sleep Apnea of Adult
MeSH Terms: interventions — Morphine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine (Active Comparator): Intrathecal Morphine 0.1mg
  Interventions: Drug: Morphine
- Fentanyl (Active Comparator): Intrathecal Fentanyl 40mcg
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Morphine — Drug: Morphine Depending on the randomization schedule, 0.1mg of morphine or will be added to the intrathecal mixture.
  Arms: Morphine
Drug: Fentanyl — Drug: Fentanyl 40mcg Depending on the randomization schedule, 40μg of fentanyl will be added to the intrathecal mixture.
  Other Names: Fentanyl-hameln
  Arms: Fentanyl

SUMMARY:
Obstructive Sleep Apnea (OSA) is a common clinical problem with a reported prevalence of 2% to 4% in the general population. The incidence was double on patients who had a diagnosis of OSA going for orthopedics surgery.

Little literature composed mostly of case reports or small retrospective case-control studies exist examining the use of intrathecal opioids on outcomes in OSA patients is inconclusive. The primary objective of this study is to compare the post operative respiratory effect after single dose intrathecal morphine and intrathecal fentanyl on orthopedics patients who suspected or undiagnosed obstructive sleep apnea.

Hypotheses

Undiagnosed OSA patients who received intrathecal morphine are more likely to have respiratory events post-operatively.

DETAILED DESCRIPTION:
This is a prospective, randomized study to compare the post operative respiratory effect after single dose intrathecal morphine (0.1mg) and intrathecal fentanyl (40mcg) on orthopedics patients who suspected or undiagnosed obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. ASA I - II
3. Patients who admitted for orthopedic surgery and consented for regional anesthesia
4. STOP - BANG score ≥ 5

Exclusion Criteria:

1. Refused to give informed consent
2. Previous diagnosis and treatment of OSA or any sleep-related breathing disorder
3. Allergic to morphine / fentanyl / Local anesthetic
4. Contra-indicated for regional anesthesia
5. Pregnant woman
6. Contraindication to either of the oral analgesia as in protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Respiratory Rate (RR) | 72 hours post operatively
  The end point of the study is to assess the respiratory rate (RR) within 72 hours post-operatively in both arms of the patients.
Heart Rate (HR) | 72 hours post-operative
  The end point of the study is to assess the heart rate (HR) within 72 hours post-operatively in both arms of the patients.
Oxygen Desaturation Index (ODI) | 72 hours post-operative
  The end point of the study is to assess the Oxygen Desaturation Index (ODI) within 72 hours post-operatively in both arms of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Chew Yin, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia